CLINICAL TRIAL: NCT06948097
Title: Syk Inhibition in MItigating Lung Allograft Rejection (SIMILAR): A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Dose Escalation Trial to Evaluate the Safety and Tolerability of Fostamatinib in Lung Transplant Patients With Donor-Specific Antibodies.
Brief Title: Syk Inhibition in MItigating Lung Allograft Rejection (SIMILAR): A Trial to Evaluate the Safety and Tolerability of Fostamatinib in Lung Transplant Patients With Donor-Specific Antibodies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10002084; 002084-H
Record Dates: First submitted 2025-04-26; First posted 2025-04-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Lung Transplantation
Keywords: Fostamatinib; Lung Transplant; Donor-specific antibodies; Antibody-mediated rejection
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fostamatinib (Experimental): Patients will receive fostamatinib with standard of care to assess safety in LT recipients with positive DSA.
  Interventions: Drug: fostamatinib
- Placebo (Placebo Comparator): Patients will receive placebo with standard of care to assess safety in LT recipients with positive DSA.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fostamatinib — The study intervention is fostamatinib, administered orally starting at 100 mg daily for 14 days, escalating to 100 mg BID for 14 days, then 150 mg BID for 28 days, based on tolerability. Patients will be monitored for 28 additional days and randomized to receive either fostamatinib or placebo, along with standard of care.
  Arms: Fostamatinib
Drug: Placebo — Placebo tablets will match fostamatinib, starting at 100 mg daily for 14 days, escalating to 100 mg BID for 14 days, and then 150 mg BID for 28 days, based on tolerability. Patients will be monitored for an additional 28 days.
  Arms: Placebo

SUMMARY:
Background:

People who have lung transplants often survive 6 or 7 years. But some people develop donor-specific antibodies (DSA) after their transplants; antibodies are proteins that attack foreign invaders in the body. Antibodies typically kill viruses and other agents that can cause disease. But when the antibodies attack a transplanted organ, they can cause the body to reject the new tissues. People who develop DSA after a transplant have a higher risk of death within 1 year.

Objective:

To test a drug called fostamatinib in people who develop DSA after a lung transplant.

Eligibility:

Adults aged 18 and older who developed DSA after a lung transplant.

Design:

Participants will continue with their standard care after a transplant.

Fostamatinib is a pill taken by mouth. Some participants will take the study drug along with their standard care; others will take a placebo. A placebo is a pill that looks just like the real drug but contains no medicine. All participants will take 1 pill per day for 2 weeks. Then they will take 2 pills per day for the next 6 weeks.

Participants will have clinic visits every 2 weeks while taking their pills. They will have a physical exam, with blood and urine tests, during each visit.

If participants have fluid samples collected from their airways during their standard treatment, some extra fluid may be collected for this study.

Participants will have a follow-up visit 4 weeks after they stop taking their pills.

DETAILED DESCRIPTION:
Study Description:

The overall objective of this study is to assess the clinical safety and tolerability of fostamatinib in lung transplant (LT) patients with positive donor-specific antibodies (DSA). Subjects who tested positive for DSA will be enrolled. Randomization to fostamatinib or placebo will be blinded. Patients will receive fostamatinib or placebo, first 100 mg orally daily for 2 weeks, then escalate to 100 mg orally twice daily for an additional 2 weeks, and then escalate to 150 mg twice daily for an additional 4 weeks. Subjects will be monitored for 28 additional days. The primary outcome is the number of discontinuations of study drug. Secondary outcomes will evaluate other safety parameters, as well as potential clinical and molecular benefits of fostamatinib in the prevention of antibody-mediated rejection (AMR) in DSA+ LT patients.

Objectives:

Primary Objective:

To assess the clinical safety and tolerability of fostamatinib compared to placebo in DSA+ LT patients.

Secondary Objectives:

To evaluate molecular and clinical benefit of fostamatinib compared to placebo in DSA+ LT patients.

Exploratory Objective:

To gain additional molecular insight into the mechanism of fostamatinib in DSA+ LT patients.

Endpoints:

Primary Endpoint:

-Incidence and relationship to study drug of the following: hypertension, neutropenia, diarrhea, increase LFTs requiring discontinuation of study drug.

Secondary Endpoints:

* Rate of DSA clearance
* Relative change of forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) from baseline to Day 56 and from baseline to Day 84
* Number of patients who has discontinued the study drug or placebo without restarting by the end of each dose (Day 14, 28, 56) due to serious adverse events
* Incidence of clinical AMR
* Number of temporal holds of study drug at different study drug dose.
* Number of patients with missed doses of study drug at each study visit.
* Number of doses missed at each study drug dose level.
* Total number of drug dose by day 56.

Exploratory Endpoints:

* Adverse events not specified in primary or secondary endpoints: incidence, severity and relationship to study drug
* Bronchoalveolar lavage (BAL) neutrophil extracellular trap (NET) production
* Plasma tissue-specific cell free (cf)DNA levels at baseline, Day 14, Day 28, Day 42, Day 56, Day 84.
* Measure blood concentration of fostamatinib at each dose. This will be measured at the end of the study to prevent unblinding.
* Relative change of molecular markers (NETs, interleukin 6, double stranded [dd]cfDNA) at baseline, Day 14, Day 28, Day 42, Day 56, and Day 84.
* Rate of DSA clearance, relative change of forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) from baseline to Day 56 and from baseline to Day 84.
* Differential gene expression from RNA sequencing of BAL fluid and PBMCs for drug and placebo
* cf DNA, cytokine, and NET at the time of clinical complication

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who do not meet any of the following criteria during screening will not be randomized but will be counted toward study accrual. Screen failures may be rescreened at a later time if the reason for screening failure is revised. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* First time LT recipients
* Have provided signed written informed consent, prior to performing any study procedure, including screening procedures.
* Age greater than or equal to 18 years
* Patients who first test positive for class II DSA between day 21 and day 180 post-transplantation, and screened within 14 days of first testing positive.
* No prior demonstration of DSA
* Demonstrate no clinical or spirometry signs of allograft dysfunction at the time of enrollment.
* Have adequate liver function, as defined by:

  * Serum aspartate aminotransferase (AST) <=1.5 x Upper Limit of Normal (ULN) (unless the increased AST is assessed by the Investigator as due to hemolysis) and alanine aminotransferase (ALT) <=1.5 x ULN.
  * Absolute neutrophil count >=1.0 x 10^9/L.
  * Hemoglobin >= 9 g/dL
* For women of reproductive potential, have a negative serum pregnancy test during the screening period. Women of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal (i.e., who have not menstruated at all for at least the preceding 1 year prior to signing informed consent unrelated to hormonal contraception).
* For women of reproductive potential, be abstinent as part of their usual lifestyle, or agree to use 2 effective forms of contraception from the time of giving informed consent, during the study, and for 28 days following the last dose of study treatment. An effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine or subdermal contraceptive implants, and barrier methods.
* Be willing to comply with all study procedures for the duration of the study.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Have a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data. Such significant medical conditions include, but are not limited to the following:

  * History of neutropenia (benign ethnic neutropenia and/or acquired neutropenia).
  * History of posterior reversible encephalopathy syndrome (PRES)
  * History of poorly controlled hypertension or hypertensive crises (defined as systolic blood pressure >=180 mmHg or average diastolic blood pressure >=120 mmHg based on an average of 3 blood pressure readings despite adequate antihypertensive therapy) unless controlled for >90 days prior to enrollment.
  * History of positive post-transplant active hepatitis C and/or hepatitis B viral infection.
  * History of drug-induced cholestatic hepatitis.
  * History of any primary malignancy, with the exception of: curatively treated nonmelanomatous skin cancer; curatively treated cervical or breast carcinoma in situ; or other primary tumor treated with curative intent, no known active disease present, and no treatment administered during the last 5 years.
  * Testing positive for human immunodeficiency virus 1 or 2 Ab with evidence for ongoing active infection (i.e., CD 4 count <400/microliter and viral load >100,000 copies/ml) on antiretroviral therapy.
  * Current or recent history of psychiatric disorder that, in the opinion of the Investigator or Medical Monitor, could compromise the ability of the subject to cooperate with study visits and procedures.
  * Are currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo.
  * Having had a prior lung or any organ transplant.
  * Currently pregnant or lactating.
  * Estimated glomerular filtration (eGFR) rate less than 30 mL/min.
  * Current or history of grade 3 diarrhea.
* Subjects on strong CYP3A4 inducers.
* Subjects who have received prior treatment for DSA.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-07-14 (Estimated); Study Completion 2028-07-14 (Estimated)

PRIMARY OUTCOMES:
Study Drug Discontinuation Rate. | 12 weeks
  The primary outcome is the number of participants who discontinue the study drug due to adverse events, intolerance, or other reasons during the treatment period.

SECONDARY OUTCOMES:
Safety and AMR Prevention in DSA+ LT Patients. | 12 weeks
  Secondary outcomes will evaluate additional safety parameters and explore the clinical and molecular benefits of fostamatinib in preventing antibody-mediated rejection (AMR) in DSA+ LT patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sean T Agbor-Enoh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (5):
- United States (5):
  - Stanford University School of Medicine, Stanford, California
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland
  - University of Utah Health, Salt Lake City, Utah
  - Inova Health System Foundation, Falls Church, Virginia